CLINICAL TRIAL: NCT06010108
Title: Actions For Collaborative Community Engaged Strategies for HPV (ACCESS-HPV)
Brief Title: Actions For Collaborative Community Engaged Strategies for HPV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Nigerian Institute of Medical Research (Other Government); University of North Carolina, Chapel Hill (Other)
Responsible Party: Principal Investigator, Juliet Iwelunmor, PhD, Professor of Medicine, Washington University School of Medicine
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NHREC/01/01/2007
Record Dates: First submitted 2023-08-07; First posted 2023-08-24 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: HPV; Stigma
MeSH Terms: conditions — Social Stigma

STUDY DESIGN:
Intervention Model Description: intervention pilot
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Heroes for Her (Active Comparator): Market outreach intervention- Community entry to engage major stakeholders. Awareness of the project will be made in the community through a public market crier who makes public announcements in the market daily using an audio recording. Lead/Mentor mothers who are mothers from the neighbourhood will be recruited to go door-to-door to reach out to the community. Before the screening and vaccination exercise, the woman will be counselled properly and taught about the HPV self-screening procedure. Mothers are expected to come to the hospital when returning their samples with their daughter so their daughter receive the vaccine
  Interventions: Behavioral: Heroes for Her
- The Reach Initiative (Active Comparator): School based intervention-The Reach Initiative involves the Mother-Daughter Day (MDD) to create awareness and provide screening and vaccination to women and girls. This will adopt the following components. MDD which is a campaign that includes educative activities and participants will be given souvenir packs containing key-cards. On-site vaccination and sample collection kits education to be provided by healthcare providers.
  To foster community engagement and promote sustainability, mothers and daughters will be encouraged to volunteer to be on the Mother-Daughter Planning Committee and participate in creating awareness.
  Interventions: Behavioral: The Reach Initiative
- W.H.I.T.E Project (Active Comparator): Community based intervention- Community engagement by consulting with stakeholders in the community, and seeking their support for the W.H.I.T.E Project through advocacy visits. Study participants will be recruited through community based outreaches and will be educated on Human Papilloma virus and cervical cancer. This will be carried out through inter-personal communication, and use of Information, Education and Communication (IEC) materials designed for the purpose of this intervention.
  Vaccination of girls age 9-14years recruited for the study will be through referral to the service point (health facility) and vaccination at outreach site.
  The W.H.I.T.E self-sample kit, will be distributed to women age 30 to 65 years through referral to the service point and distribution at outreach site.
  Interventions: Behavioral: W.H.I.T.E project
- Project Shield (Active Comparator): Distribution of branded self-sampling kits for HPV screening and vaccination through community based structures- Participants will be recruited through fliers, posters and community volunteers. The branded kit will include the Evalyn brush, sanitary pad/panty liner, a user manual which will be translated in local languages. Mothers who purchase the self-sampling kit will receive a free vaccination voucher for their daughters. The kits will be sold at a discounted rate. The voucher will enable the daughters to receive the HPV vaccine for free. To create awareness about cervical cancer, banners will be displayed at pharmacies and the community health facilities. The Community Development Association (CDA) will participate in awareness campaigns utilizing local languages and culturally appropriate messages. Community hospitals and pharmacies will serve as points of access for the self-sampling kits and vaccines.
  Interventions: Behavioral: Project Shield
- Project SHADE (Active Comparator): Community based intervention using a uniquely designed bag "Eno Iban" to package and distribute the self collection kit and use of a simple app (d-SHADE) to collect participants data- Community outreaches will be carried out in several areas within the community such as markets to create awareness on cervical cancer prevention and to recruit women and girls. Female healthcare providers will be actively involved in these outreaches. Interested participants will be given uniquely branded kits containing a self-sampling brush from the mothers and a vaccination voucher for daughters. Mothers will be required to collect their samples either at the community facility or at home. When returning the Samples to the community facility, mothers will be expected to come with their daughters who then receive the HPV vaccination. All collected samples will be returned to the reference laboratory for analysis
  Interventions: Behavioral: Project SHADE
- Operation Reach Her (ORH) (Active Comparator): Faith-based intervention- Reaching women and girls through places of religious worship and religious leaders. Awareness programs would be conducted in the chosen religious centres to educate women and girls about their health, cervical cancer, its prevention. This would be achieved by organizing a " Health Day " for free health check-ups for all members of the congregation. HPV screening and vaccination would be a part of these check-ups. Announcements would be carried out in worship centres to enrol women and girls. HPV vaccination to girls will be provided by health care providers stationed at the religious centres in the area. The self-sampling kit would be distributed to women in mobile tents stationed in churches and mosques. Girls who have been successfully vaccinated would receive a vaccination card and wristband to show that they have been vaccinated. The self-sampling kits would be collected from the women on the same day and transported to the reference laboratory
  Interventions: Behavioral: Operation Reach Her (ORH) program
- Project Care (Active Comparator): Use of community pharmacies to promote awareness and serve as service points for self-collection and vaccination-Trained pharmacists and healthcare workers, student pharmacists, and students in other fields of study will serve as ambassadors to recruit, provide education and provide guidance on the use of the self- sample kit when needed. Participants will be recruited through community outreach programs, awareness campaigns in hair saloons, workplaces, social media and collaboration with local healthcare facilities. In addition, pharmacies will display promotional materials and provide information to potential participants. Dedicated areas within the local pharmacies will be set up for screening and vaccinations. The mothers and daughters on participation will be given hair accessories as incentives. The screening and HPV vaccination will also be provided at discounted prices.
  Interventions: Behavioral: Project Care

INTERVENTIONS:
Behavioral: Heroes for Her — Market outreach intervention- daily awareness creation through public market announcements, and distribution of educational fliers in local dialects. Community women will also be involved in the spread awareness through door to door approach. Thee will be repeated radio jingles to promote awareness. Interested women and girls will be provided with screening and vaccination services at a designated community health facility. All samples will be returned to the facility by the women and sent to a designated laboratory for testing. Participants contact information will be collected for follow up
  Arms: Heroes for Her
Behavioral: The Reach Initiative — School based intervention-The Reach Initiative involves the organisation of the Mother-Daughter Day (MDD) by Mother-Daughter Planning Committee (MDPC) who are volunteer young school girls and their mothers and provision of a Key-Card which is a cervical cancer awareness card attached to a key chain for awareness creation. HPV vaccination and HPV -self sampling will be carried out in private rooms within the venue of the intervention and all samples will be sent to designated laboratory for testing. Participants contact information will be collected for follow up and communication of results
  Arms: The Reach Initiative
Behavioral: W.H.I.T.E project — Community based intervention- This will involve the engagement of women's trade unions and organisations in the community to create awareness and women and girls interested in the uptake of HPV prevention services will be directed to receive these services at a designated community facility accessible to women and girls in the community. Participants contact details will be collected for follow uo and communication of results
  Arms: W.H.I.T.E Project
Behavioral: Project Shield — Utilization of community based structures (pharmacy and health center)- The intervention will involve the creation of a branded self-sampling kit for HPV screening and a free vaccination voucher to encourage mother-daughter uptake of cervical cancer prevention measures. Awareness will be raised through banners at the points of access of the vaccines and kits, use of jingles, and the involvement of the Community Development Association (CDA) to help mobilize girls, women and the men. Women and girls will be referred to community health centers to receive the HPV vaccination and carry out the screening
  Arms: Project Shield
Behavioral: Project SHADE — Community-based approach- health education of girls and women. The use of a uniquely designed bag "Eno Iban" to package and distribute the self-collection tool, vaccination of the adolescent girls. Screening and HPV will be provided at designated areas within the community for women and girls. A simple app (d-SHADE) will be used to collect data of the girls and women by the health professionals and volunteers, as well as send the reminders for next screening dates and test results
  Arms: Project SHADE
Behavioral: Operation Reach Her (ORH) program — Faith based approach- Awareness programs would be conducted in the chosen religious centres to educate women and girls about their health, cervical cancer, its prevention, and the benefits of screening and HPV vaccination. This would be achieved by organizing a " Health Day " for free health check-ups for all members of the congregation. The self-sampling kit would be distributed to women aged 30-65 in mobile tents stationed in churches in Akoka and HPV vaccinations would be administered to girls aged 9-14 in mobile tents stationed at churches and mosques in Akoka, Lagos
  Arms: Operation Reach Her (ORH)
Behavioral: Project Care — Community pharmacy intervention-Trained community volunteers will be involved in creating awareness of HPV prevention services and cervical cancer. There will be distribution of cervical cancer self-sampling kits to community pharmacies which will serve as service points for screening (self-collection point) and vaccination point for girls in the community,
  Arms: Project Care

SUMMARY:
In the current pilot study, Actions for Collaborative Community-Engaged Strategies for HPV (ACCESS-HPV), investigators will use participatory crowdsourcing methods to drive HPV prevention among mother-daughter dyads. Crowdsourcing open calls will allow us to identify locally relevant messages and dissemination techniques to increase uptake of HPV prevention. Then, participatory learning communities will build capacity for community led implementation of selected strategies. Informed by social learning theory and the PEN-3 cultural model, our multi-disciplinary research team proposes the following specific aims: (1) to develop a new combined campaign to increase HPV vaccination for young girls (ages 9-14) and HPV self-collection for mothers (ages 30-65) using crowdsourcing open calls and participatory learning communities; and (2) to determine the preliminary effectiveness of, seven crowdsourced campaign on uptake of HPV vaccination among young girls/women and HPV self-collection among their mothers. Our primary outcome will be HPV vaccine uptake (ascertained by clinic records of vaccine uptake) among young girls and HPV self-collection (ascertained by laboratory receipt of specimens) among their mothers. The strong support of the Nigerian Institute for Medical Research (NIMR) alongside national HPV programs creates a rich research infrastructure and increases the likelihood of successful implementation. Our multi-disciplinary research team has experience organizing implementation research focused on crowdsourcing and community participation in Nigeria. This pilot study will enhance our understanding of HPV prevention in resource-constrained settings.

DETAILED DESCRIPTION:
Step 1: Health facilities training. For the purposes of this research study, the Nigerian Institute of Medical Research team would provide training to health centers currently working with the Nigerian Institute of Medical Research .The training would be to ensure that these health facilities are trained to provide follow up services to participants who be referred. Following the training, the NIMR research team would in charge of collecting data to record participants HPV self-collection uptake and HPV vaccination uptake.

Step 2: Participant enrollment. This will involve recruiting women and girls to participate in the pilot study. Participant recruitment strategies will include: social media, online, event- and venue based, participant referral, and walk-ins at study clinics. Participant enrollment will be completed by study team.

Step 3: Baseline data collection. After enrollment, study team will collect baseline data on HPV self-collection and cervical cancer screening history, knowledge of cervical cancer, HPV screening, determine the role of intersectional stigma on barriers and facilitators of HPV-related service delivery (HPV vaccination/HPV self-collection) among Nigerian girls and women, assess the feasibility, acceptability, and preliminary impact of three asset-based mother-daughter interventions that address intersectional stigma and HPV service uptake among Nigerian girls and women and other related outcomes will be collected from recruited participants. Participants mobile phone numbers will also be collected as tracking information for follow-up and retention in a coupon format. The mobile phone numbers would be used to contact study participants through text messages and phone calls. These contacts would serve as reminders for participants to participate in follow-up data collection. The mobile phone service charge would be covered by the research. No other personal identifiers will be collected and no biological specimens will be collected at baseline. The investigators will obtain informed consent before proceeding with any data collection.

Step 4: Intervention implementation. Following participant recruitment and enrollment in the study as well as completion of baseline study, participants will be assigned to one of the seven mother-daughter interventions focused on expanding the uptake of HPV self-sampling, HPV vaccination and addressing stigma associated with HPV prevention services uptake among Nigerian women and girls.The pilot intervention implementation would occur for 30 days. Nigerian Institute of Medical Research (NMIR) will provide local training on HPV prevention to the seven participatory interventions following their existing guidelines. The participatory interventions will be conducted in the locations of the seven teams who emerged as winners from the innovation boot-camp. These participatory interventions will only provide HPV self-sampling and vaccination and instructions of how to perform the test to participants. They will also provide referral coupons to women who test positive or participants who have any adverse effects. The referral coupons are intended to provide study participants information on health facilities and specialists that are involved with the research. The intervention only provide participants with the HPV self-collection and vaccination kits and does not involve monitoring HPV self-collection procedure, the investigators will only be asking for self-reported HPV self-collection and vaccination uptake

Step 5: Follow up surveys at 8 weeks. At 8 weeks post intervention implementation, study team will collect similar baseline data from study participants. The follow-up survey will assess HPV self-testing, HPV vaccination assess the feasibility, acceptability, and preliminary impact of 7 mother-daughter interventions focused on expanding the uptake of HPV self-sampling, HPV vaccination and addressing stigma associated with HPV prevention services uptake among Nigerian women and girls.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Both the mothers'/caregivers' (between ages 30-65 years) and daughters' (Between 9 to 14 years) willingness to participate in the study
* All participants must agree to an informed consent in English
* Parental guardian's cell phone number for follow-up and/or retention

Exclusion Criteria:

Inability to comply with study protocol

* Illness, cognitive impairment or threatening behavior with acute risk to self or others
* No informed consent or cell phone

Ages: 9 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 350 (Actual)
Dates: Start 2024-01-15 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
Uptake of HPV Vaccination Over the 8 weeks follow-up | 8 weeks following the first encounter
  Proportion of eligible girls who receive at least one dose of HPV vaccine at 8 weeks after baseline. This will be ascertained by clinic records of vaccine uptake.
Uptake of HPV Self-collection Over the 8 weeks Follow-up | 8 weeks following the first encounter
  Proportion of eligible women who complete an HPV self-test at 8 weeks after baseline. This will be ascertained by laboratory receipt of self-collected specimens.

SECONDARY OUTCOMES:
Intersectional Discrimination Index | Measured at baseline and at 8 weeks
  HPV-and-cervical cancer associated stigma will be assessed using the Intersectional Discrimination Index measure. Higher scores mean greater stigma.
Intervention Acceptability | Measured at baseline and at 8 weeks
  This will be assessed using the Acceptability of Intervention Measure (AIM). The subscale is rated on a 5-point Likert scale, 1 to 5 with higher scores indicating higher levels of acceptability.
Intervention Appropriateness | Measured at baseline and at 8 weeks
  This will be assessed using the Intervention Appropriateness Measure (IAM). The subscale is rated on a 5-point Likert scale, 1 to 5 with higher scores indicating higher levels of Appropriateness.
Intervention Feasibility | Measured at baseline and at 8 weeks
  This will be assessed using the Feasibility of Intervention Measure (FIM). The subscale is rated on a 5-point Likert scale, 1 to 5 with higher scores indicating higher levels of feasibility.

OTHER OUTCOMES:
Key Implementation Factors | Up to 8 weeks
  Guided by the RE-AIM framework for implementation science, semi-structured, in-depth interviews will be conducted at the individual and setting levels to explore the factors associated with the implementation of the intervention (e.g., reach, adoption, implementation, and maintenance).

CONTACTS AND LOCATIONS:
Locations (1):
- Nigerian Institute of Medical Research, Yaba, Lagos, Nigeria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Campos NG, Demarco M, Bruni L, Desai KT, Gage JC, Adebamowo SN, de Sanjose S, Kim JJ, Schiffman M. A proposed new generation of evidence-based microsimulation models to inform global control of cervical cancer. Prev Med. 2021 Mar;144:106438. doi: 10.1016/j.ypmed.2021.106438. Epub 2021 Mar 4. PMID 33678235
- [Background] McFarland DM, Gueldner SM, Mogobe KD. Integrated Review of Barriers to Cervical Cancer Screening in Sub-Saharan Africa. J Nurs Scholarsh. 2016 Sep;48(5):490-8. doi: 10.1111/jnu.12232. Epub 2016 Jul 19. PMID 27434871
- [Background] Lim JN, Ojo AA. Barriers to utilisation of cervical cancer screening in Sub Sahara Africa: a systematic review. Eur J Cancer Care (Engl). 2017 Jan;26(1). doi: 10.1111/ecc.12444. Epub 2016 Feb 7. PMID 26853214
- [Background] Devarapalli P, Labani S, Nagarjuna N, Panchal P, Asthana S. Barriers affecting uptake of cervical cancer screening in low and middle income countries: A systematic review. Indian J Cancer. 2018 Oct-Dec;55(4):318-326. doi: 10.4103/ijc.IJC_253_18. PMID 30829264
- [Background] Amponsah-Dacosta E, Kagina BM, Olivier J. Health systems constraints and facilitators of human papillomavirus immunization programmes in sub-Saharan Africa: a systematic review. Health Policy Plan. 2020 Jul 1;35(6):701-717. doi: 10.1093/heapol/czaa017. PMID 32538437
- [Background] Abuelo CE, Levinson KL, Salmeron J, Sologuren CV, Fernandez MJ, Belinson JL. The Peru Cervical Cancer Screening Study (PERCAPS): the design and implementation of a mother/daughter screen, treat, and vaccinate program in the Peruvian jungle. J Community Health. 2014 Jun;39(3):409-15. doi: 10.1007/s10900-013-9786-6. PMID 24276617
- [Background] Winer RL, Gonzales AA, Noonan CJ, Buchwald DS. A Cluster-Randomized Trial to Evaluate a Mother-Daughter Dyadic Educational Intervention for Increasing HPV Vaccination Coverage in American Indian Girls. J Community Health. 2016 Apr;41(2):274-81. doi: 10.1007/s10900-015-0093-2. PMID 26399648
- [Background] Scarinci IC, Hansen B, Kim YI. HPV vaccine uptake among daughters of Latinx immigrant mothers: Findings from a cluster randomized controlled trial of a community-based, culturally relevant intervention. Vaccine. 2020 May 22;38(25):4125-4134. doi: 10.1016/j.vaccine.2020.03.052. Epub 2020 Apr 27. PMID 32354671
- [Background] Lee H, Kim M, Cooley ME, Kiang PN, Kim D, Tang S, Shi L, Thiem L, Kan P, Peou S, Touch C, Chea P, Allison J. Using narrative intervention for HPV vaccine behavior change among Khmer mothers and daughters: A pilot RCT to examine feasibility, acceptability, and preliminary effectiveness. Appl Nurs Res. 2018 Apr;40:51-60. doi: 10.1016/j.apnr.2017.12.008. Epub 2017 Dec 18. PMID 29579499
- [Background] Cates JR, Shafer A, Diehl SJ, Deal AM. Evaluating a County-Sponsored Social Marketing Campaign to Increase Mothers' Initiation of HPV Vaccine for their Pre-teen Daughters in a Primarily Rural Area. Soc Mar Q. 2011 Spring;17(1):4-26. doi: 10.1080/15245004.2010.546943. PMID 21804767
- See also: Global strategy to accelerate the elimination of cervical cancer as a public health problem — http://www.who.int/publications/i/item/9789240014107